CLINICAL TRIAL: NCT06448299
Title: Erector Spinae Plane Block Versus Oblique-Subcostal Transversus Abdominis Plane Block in Patients Undergoing Emergency Abdominal Surgery with Midline Incision: a Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Oblique-Subcostal Transversus Abdominis Plane Block in Emergency Abdominal Surgery with Midline Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-305-2023
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative; Abdominal Surgery; Emergency
MeSH Terms: conditions — Pain, Postoperative; Emergencies | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAPB (Active Comparator)
  Interventions: Procedure: TAPB
- ESPB (Active Comparator)
  Interventions: Biological: ESPB

INTERVENTIONS:
Procedure: TAPB — Patients will receive ultrasound guided bilateral oblique subcostal TAPB using 25 mL bupivacaine 0.25% in each side
  Arms: TAPB
Biological: ESPB — Patients will receive ultrasound guided bilateral ESPB at T8 level using 25 mL bupivacaine 0.25% in each side
  Arms: ESPB

SUMMARY:
Most of the recommendations regarding pain management in emergency abdominal surgery are extracted from data from elective abdominal surgery. However, surgery in the emergency settings differs from the elective settings in the extent stress and the pain which is usually present preoperatively; therefore, it is expected to have different analgesic requirements and different response to pain management interventions in emergency surgery.

Abdominal wall blocks are increasingly used in abdominal surgery. However, data regarding their efficacy in emergency setting are lacking. Oblique-subcostal transversus abdominis plane block (OS-TAPB) is a variation of the subcostal TAPB that could achieve effective analgesia for both upper and lower parts of the abdomen. The TAPB characterized by being easy to perform and does not require patient repositioning. Erector spinae plane block (ESPB) is another abdominal wall block that showed good analgesic effect following various elective open abdominal surgeries, but the block requires patient repositioning before block performance. In elective abdominal surgeries, the current evidence slightly supports ESPB over the TAPB. We hypothesize that the difference between the two blocks would be more apparent in in emergency surgery due to the type of incision, extent of tissue manipulation, and severity of pain.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and pre-medication drugs will be delivered (metoclopramide 10 mg and omeprazole 40 mg).

General anesthesia will be induced by 2 mg/kg propofol and 1 mcg/kg fentanyl. After loss of consciousness, tracheal intubation by direct laryngoscopy will be facilitated by 1 mg/kg succinyl choline. Anesthesia will be maintained by 1-1.2% isoflurane and atracurium will be administered after patient recovery from succinylcholine at a dose of 0.5 mg/Kg. Atracurium increments of 0.1 mg/kg will be administered every 20 min for maintenance of neuromuscular blockade.

After induction of anesthesia, patients will receive the block according to the group assignment In both blocks a total of 25 mL of 0.25% bupivacaine will be administered in each side.

The blocks will be performed by an experienced operator who will be informed of the patient group after induction of anesthesia. The patient, surgeon and data collector will be blinded to the study group.

Intraoperative analgesic management Fentanyl boluses of 1 mcg/kg will be given in case of inadequate analgesia (heart rate/mean blood pressure increase by 20% from the baseline in absence of other causes) Intraoperative fluid and hemodynamic management will be according to the discretion of the attending anesthetist.

At the end of the surgery, all patients will receive intravenous acetaminophen (1 g) before the extubation.

Postoperative care All patients will receive regular intravenous acetaminophen 1 g/6 hours. Pain assessments using NRS will be performed at rest and during cough at 0.5, 1, 4, 8, 12, 24 h after leaving the operating room. If NRS score is > 3 (at any time not limited to the time of assessment) intravenous titration of 3 mg morphine is given slowly to be repeated after 30 minutes if pain persisted. If other opioids are given, morphine equivalent dose will be calculated using opioids conversion chart.

Intravenous ondansetron 4 mg will be given to treat nausea or vomiting if occurs

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years), undergoing emergency abdominal surgery with midline incision

Exclusion Criteria:

* American society of anesthesiologist-physical status >III,
* patients with a history of allergy to any of the study drugs,
* a body mass index (BMI) <18 or ≥ 40 kg/m2,
* coagulopathy
* local infection,
* history of chronic pain or regular opioid use;
* inability to comprehend the Numeric Rating Scale (NRS),
* pregnant or lactating women. Patients on vasopressor infusion,
* patients with high shock index (heart rate / systolic blood pressure >1)
* patients requiring postoperative mechanical ventilation will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption | 30 minutes postoperatively till 24 hours postoperatively
  mg

SECONDARY OUTCOMES:
numerical rating scale at rest | 30 minutes postoperatively till 24 hours postoperatively
  11-points scale in which the patients are asked to circle the number between 0 and 10 that best describe their pain intensity. Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible) will be performed at rest and during cough at 0.5, 1, 4, 8, 12, 24 h after leaving the operating room
numerical rating scale during cough | 30 minutes postoperatively till 24 hours postoperatively
  11-points scale in which the patients are asked to circle the number between 0 and 10 that best describe their pain intensity. Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible) will be performed at rest and during cough at 0.5, 1, 4, 8, 12, 24 h after leaving the operating room
Time to first morphine requirement | 30 minutes postoperatively till 24 hours postoperatively
  hours
Time to independent movement | 30 minutes postoperatively till 24 hours postoperatively
  hours
postoperative sedation | 30 minutes postoperatively till 24 hours postoperatively
  modified Ramsay Sedation score
patients satisfaction | 24 hours postoperatively
  using the NRS 0= worst experience, 10= best experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data related to this study will be provided from the PI upon reasonable request